CLINICAL TRIAL: NCT03309332
Title: OSB Lead-AMPLATZER PFO Occluder New Enrollment PAS
Brief Title: AMPLATZER PFO Occluder Post Approval Study
Acronym: PFO PAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SJM-CIP-10187
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Patent Foramen Ovale
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device (Experimental): Subjects implanted with the AMPLATZER™ PFO Occluder.
  Interventions: Device: AMPLATZER™ PFO Occluder

INTERVENTIONS:
Device: AMPLATZER™ PFO Occluder — Implantation of the AMPLATZER™ PFO Occluder in the PFO

SUMMARY:
The purpose of this single arm, multi-center study is to confirm the safety and effectiveness of the AMPLATZER™ PFO Occluder in the post Approval Setting.

DETAILED DESCRIPTION:
A maximum of 1214 adult subjects will be enrolled at up to 100 centers in the U.S. and Canada. Subjects will have follow-up at 1 month, 6 months, 12 months and annually thereafter through 5 years post implant.

ELIGIBILITY:
Inclusion Criteria:

• Subjects with a PFO who have had an ischemic stroke within the last 547 days

Exclusion Criteria:

* Atherosclerosis or other arteriopathy of the intracranial and extracranial vessels associated with a ≥ 50% lumen diameter supplying the involved lesion
* Intra-cardiac thrombus or tumor
* Documented evidence of venous thrombus in the vessels through which access to the PFO is gained
* Acute or recent (within 6 months prior to consent) myocardial infarction or unstable angina
* Left ventricular aneurysm or akinesis
* Mitral valve stenosis or severe mitral regurgitation requiring intervention irrespective of etiology
* Aortic valve stenosis (mean gradient >40 mmHg) or severe aortic valve regurgitation
* Mitral or aortic valve vegetation or prosthesis
* Aortic arch plaques protruding greater than 4mm into the aortic lumen
* Left ventricular dilated cardiomyopathy with depressed left ventricular ejection fraction (LVEF less than 35%)
* Subjects with other source of right to left shunts, including an atrial septal defect and/or fenestrated septum
* Chronic, persistent, or paroxysmal atrial fibrillation or atrial flutter
* Pregnancy at the time of implant
* Age less than 18 years or greater than 60 years at time of consent
* Active endocarditis or other untreated infections
* Organ failure (kidney, liver or lung). Kidney failure: Poor urine output of less than 1 cc/kg/hr with elevated BUN levels (above the normal reference range for the laboratory at the investigational site). Liver failure: Liver enzymes outside the normal reference range for the laboratory at the investigational site: poor liver function as assessed by elevated PT (above the normal reference range for the laboratory at the investigational site) and low total protein and albumin (below the normal reference range for the laboratory at the investigational site). Lung failure: Respiratory failure is retention of carbon dioxide more than 60 mmHg, poor oxygenation with oxygen tension less than 40 mmHg in room air or the need for assisted ventilation.
* Uncontrolled hypertension defined as sustained elevated systemic blood pressure to more than 160/90 mmHg with medications
* Uncontrolled diabetes defined as continued elevated glucose levels in spite of administration of insulin/levels of more than 200 mg with presence of glucose in the urine
* Diagnosis of lacunar infarct probably due to intrinsic small vessel as qualifying stroke event Definition: Ischemic stroke in the distribution of a single, small deep penetrating vessel in a patient with any of the following: 1) a history of hypertension (except in the first week post stroke); 2) history of diabetes mellitus; 3) Age >/= 50; or 4) MRI or CT shows leukoaraiosis greater than symmetric, well-defined periventricular caps or bands (European Task Force on Age-Related White Matter Changes rating scale score > 0)
* Arterial dissection as cause of stroke
* Subjects who test positive with one of the following hypercoagulable states; Anticardiolipin Ab of the IgG or IgM (≥30), Lupus anticoagulant, B2-glycoprotein-1 antibodies (≥30) or persistently elevated homocysteine (>20)
* Unable to take antiplatelet therapy
* Anatomy in which the AMPLATZERTM PFO Occluder device size required would interfere with intracardiac or intravascular structures such as valves or pulmonary veins
* Vasculature, through which access to the PFO is gained, is inadequate to accommodate the appropriate sheath size
* Malignancy or other illness where life expectancy is less than 2 years
* Subjects who will not be available for follow-up for the duration of the trial
* Inability to obtain Informed Consent from patient
* Index stroke of poor outcome (modified Rankin score greater than 3)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1214 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2030-02-05 (Estimated); Study Completion 2030-02-05 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness: 5 year rate of recurrent ischemic stroke | Through 5 years
  5 year rate of recurrent ischemic stroke
Primary Safety: Device or procedure related serious adverse events | Through 30 days post implant
  Device or procedure related serious adverse events through 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, PhD, Study Director — Abbott
Locations (88):
- United States (78):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Scottsdale Healthcare Shea, Scottsdale, Arizona
  - Pima Heart Physicians, PC, Tucson, Arizona
  - UAMS Medical Center, Little Rock, Arkansas
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - USC University Hospital, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Sutter Medical Center, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - University of Colorado Hospital, Aurora, Colorado
  - Memorial Hospital of Colorado Springs, Colorado Springs, Colorado
  - Denver Heart, Denver, Colorado
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Augusta University, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - HCA Midwest Division, Menorah Medical Center, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Baptist Hospital East, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - McLaren Health Care Corporation, Auburn Hills, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - St. Mary's Hospital, Duluth, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Providence St. Patrick Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mount Sinai Hospital, New York, New York
  - New York Presbyterian Hospital/ Cornell University, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Novant Health Heart and Vascular Research, Charlotte, North Carolina
  - Moses H Cone Memorial Hospital, Greensboro, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Jewish Hospital, Cincinnati, Ohio
  - TriHealth Bethesda North Hospital, Cincinnati, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Mt Carmel East, Columbus, Ohio
  - Kaiser Sunnyside Medical Center, Clackamas, Oregon
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - Lexington Medical Center, West Columbia, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Ascension Texas Cardiovascular Research, Austin, Texas
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor Scott & White - The Heart Hospital Baylor Plano, Plano, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center - Heart & Vascular, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin
  - Aurora Medical Group, Milwaukee, Wisconsin
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
- Germany (2):
  - TUM Klinikum - Deutsches Herzzentrum München, München, Bavaria
  - Deutsches Herzzentrum Berlin, Berlin, State of Berlin
- Centro Cardiologico Monzino, Milan, Lombard, Italy
- Santa Maria Hospital, Lisbon, Lisbon District, Portugal
- Kantonsspital St.Gallen, Sankt Gallen, Stgalln, Switzerland
- St. Thomas Hospital, London, London, United Kingdom